CLINICAL TRIAL: NCT01146769
Title: Early Pelvic Floor Muscle Training Improves Pelvic Floor Muscle Strength in Patient After Low Anterior Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kwong Wah Hospital (Other)
Responsible Party: LAU Patrick YY, Department of Surgery, Kwong Wah Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMTIMS-01
Record Dates: First submitted 2010-06-15; First posted 2010-06-22 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2010-04

CONDITIONS: Cancer of Rectum
Keywords: Cancer of rectum; Physiotherapy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pelvic floor exercise (Experimental)
  Interventions: Other: Pelvic floor exercise
- Control (No Intervention)

INTERVENTIONS:
Other: Pelvic floor exercise — Pelvic floor strengthening exercise
  Arms: Pelvic floor exercise

SUMMARY:
The aim of study is to investigate the difference in Maximum Squeeze Pressure in patients with and without pelvic floor muscle training in low anterior resection in peri-operative period

DETAILED DESCRIPTION:
The functional outcome after low anterior resection varies greatly. Proportion of patient suffers from urgency and incontinence. Pelvic muscle disuse with atrophy and fibrosis may be a cause for the poor function. Peri-operative pelvic floor muscle training may preserve pelvic floor muscle bulk and function and thus improve functional outcome after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo low anterior resection of rectum
* Patient consented for study

Exclusion Criteria:

* Patient unable to understand pelvic floor exercise
* Patient who underwent alternative procedure
* Patient who suffers anastomotic complications after surgery
* Patient who ileostomy not closed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-10 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Maximum Squeeze Pressure | 1 week before operation and 3 months after operation

SECONDARY OUTCOMES:
Functional Outcomes | 1 week before operation and 3 months post operation
  Bowel frequency, Fecal incontinence score

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Y LAU, Principal Investigator — Department of Surgery, Kwong Wah Hospital
Locations (1):
- Department of Surgery, Kwong Wah Hospital, Hong Kong, Hong Kong